CLINICAL TRIAL: NCT03261557
Title: Cognitive Behavioral Social Skills Training in Early-onset Psychosis: Efficacy in Psychotic Symptoms, Psyshosocial Functioning and Neurobiological and Epigenetic Stress Markers.
Brief Title: Cognitive Behavioral Social Skills Training in Early Onset Psychosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Olga Puig, Clinical psychologist, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DN040595
Record Dates: First submitted 2017-08-23; First posted 2017-08-25 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Psychosis NOS
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Mental Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT + SST (Experimental): The treatment group will receive the intervention according to the CBSST protocol, adapted to adolescents.
  Interventions: Behavioral: CBT + SST
- Psychoeducation, habits and healthy lifestyle (Active Comparator): The control group will receive 3 modules intervention: psychoeducation, habits and healthy lifestyle.
  Interventions: Behavioral: Psychoeducation, habits and healthy lifestyle

INTERVENTIONS:
Behavioral: CBT + SST — It will consist of 1 individual sessions and 15 weekly periodicity group sessions distributed in 3 modules: cognitive skills module, which includes the basic principles of CBT for psychosis; Social skills module, which includes the usual strategies in HHSS training; and problem solving module.
  All patients will receive pharmacological treatment and will be followed up by their referral psychiatrist habitual.
  Arms: CBT + SST
Behavioral: Psychoeducation, habits and healthy lifestyle — Patients randomized to the control treatment will receive the same number of Individual and group sessions, with the same periodicity and format: 1 individual sessions and 15 weekly periodicity group sessions distributed in 3 modules: psychoeducation, habits and healthy lifestyle.
  All patients will receive pharmacological treatment and will be followed up by their referral psychiatrist habitual.
  Arms: Psychoeducation, habits and healthy lifestyle

SUMMARY:
Cognitive-behavioral therapy (CBT) and social skills training (SST) are recommended psychological interventions to improve symptomatology and functional recovery in psychosis. In addition, CBT may reduce hyperactivation of the brain structures responsible for the stress response. In patients with early onset psychotic disorder (EOP) there are not any previous controlled study that has analyzed the efficacy of this type of intervention.

The aim of this study is to investigate efficacy of CBT + SST in symptomatic and functional improvement after the treatment in patients with EOP. The study will also examine the potential effect of the intervention on neurobiological stress markers.

DETAILED DESCRIPTION:
Early-onset of psychotic disorders (EOP), and especially Schizophrenia, is associated with a worse clinical and psychosocial evolution than in the adult form of the illness. In the case of patients with EOP, international and national clinical guidelines recommend the combination of pharmacological treatment with CBT. However there are not any previous controlled study that has analyzed the efficacy of this type of psychological intervention.

A controlled randomized study will be carry out of CBT + SST intervention compared to a control intervention of the same duration, format and contact with a therapist. The sample will be 30 participants with a diagnosis of schizophrenia, Schizoaffective disorder or psychotic disorder not otherwise specified diagnosed between 9 and 18 years. Patiens have to be in the early phase of the disease (first 5 years after the onset) and in non-acute treatment. All participants will be evaluated before and after the intervention with clinical scales, neuropsychological battery and blood test(...). 20 healthy subjects paired by age, puberal stage and sex will be also recruited and evaluated only at baseline point. The evaluations will be carried out by blind evaluators. Intention-to-treat analysis will be carry out using the statistical package SPSS v 20.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of non-affective psychotic disorder diagnosed between age of 9 and 18 (Schizophrenia, schizoaffective disorder or psychotic disorder not otherwise specified according to DSM-V criteria).
* Critical period after the first psychotic episode (which covers the first 5 years) and in non-acute treatment

Exclusion Criteria:

* IQ <70
* Toxic dependence comorbid disorder
* Presence of Neurological disorder.

Ages: 12 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-02-22 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Psychosocial functioning | 15 weeks
  Change from baseline in social functioning questionnaires
Clinical symptoms | 15 weeks
  Change from baseline in Clinical scales

SECONDARY OUTCOMES:
Biological stress markers | 15 weeks
  Change pre-post interventionbiological stress markers registered by blood analyses
Subjective stress | 15 weeks
  Change pre-post intervention in questionnaires of perceived stress

CONTACTS AND LOCATIONS:
Overall Officials: Olga Puig, PhD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Department of Child and Adolescent Pyshicatry and Psychology, Barcelona, Catalonia, Spain